CLINICAL TRIAL: NCT01972295
Title: Registry on WATCHMAN Outcomes in Real-Life Utilization WASP Registry
Acronym: WASP
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 90879496
Record Dates: First submitted 2013-10-24; First posted 2013-10-30 (Estimated); Last update posted 2019-08-21 (Actual); Status verified 2017-06

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
This is an observational, prospective, non-randomized, multicenter study with the following objectives: (1) to compile real-world clinical outcomes data for WATCHMAN Left Atrial Appendage Closure Technology in patients who are implanted with the WATCHMAN device in a commercial clinical setting and (2) to collect health care usage data that may be needed for reimbursement of WATCHMAN technology in certain countries.

DETAILED DESCRIPTION:
Approximately 200 subjects will be enrolled in the study. Up to 10 sites in the Asia Pacific and Middle East regions will participate.

Primary analyses may include, but will not be limited to, the following: procedural complications, incidence of stroke and death. Descriptive statistics will be used for baseline, procedure and follow-up data collected through the study.

Each patient will be followed for a period of two years after implant according to the schedule and standard practice at the enrolling centers. There will be no additional visits, nor procedures, for subjects who participate in the study. Subjects are expected to be followed at implant, then at one post-implant visit (typically between 1-3 months of implant), and then annually through 2 years post implant. An intermediate visit may be scheduled in a number of patients, per physician discretion. In order to reliably capture patient status at study end, a follow-up window of 24 +/- 3 months will be considered acceptable for scheduling the last visit. For subjects who are not scheduled to visit the clinical for a follow-up, a subject contact (e.g. phone call) will ensure capture of the endpoint related information; however, it is recommended to perform an in-office visit for at least the first annual visit.

Enrollment is expected to be completed in 21 months; therefore the total study duration is estimated to be 48 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are eligible for a WATCHMAN device according to current international and local guidelines (and future revisions) and per physician discretion;
* Patients who are willing and capable of providing informed consent, participating in all testing associated with this clinical investigation at an approved clinical investigational center;
* Patients whose age is 18 years or above, or of legal age to give informed consent specific to state and national law.

Exclusion Criteria:

* Patients who are currently enrolled in another investigational study or registry that would directly interfere with the current study, except when the patient is participating in a mandatory governmental registry, or a purely observational registry with no associated treatments. Each instance should be brought to the attention of the sponsor to determine eligibility.
* Women of childbearing potential who are, or plan to become, pregnant during the time of the study (method of assessment upon physician's discretion);
* The subject is unable or not willing to complete follow-up visits and examination for the duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non-valvular atrial fibrillation
Sampling Method: Non-Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2014-01-13 (Actual); Primary Completion 2018-01-23 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Procedural complications, Stroke and Death | at implant and 2 year follow up
  Descriptive statistics will be used for baseline, procedure and follow-up data collected through the study.

CONTACTS AND LOCATIONS:
Overall Officials: Lynnett Voshage-Stahl, Study Director — Boston Scientific Corporation
Locations (9):
- Australia (3):
  - Royal Adelaide Hospital, Adelaide
  - Greenslopes, Brisbane
  - Monash Medical, Melbourne
- Queen Elizabeth Hospital, Hong Kong, Hong Kong
- Medistra Hospital, Jakarta, Indonesia
- Institut Jantung Negara, Kuala Lumpur, Malaysia
- Prince Sultan Cardiac Center, Riyadh, Saudi Arabia
- Severance Hospital, Seoul, South Korea
- Ramathibodi Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided